CLINICAL TRIAL: NCT03254888
Title: Identification of Novel Autophagy Markers in Bladder Cancer Patients
Brief Title: Autophagy Bladder Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shaimaa Ramadan, Principal investigator, Assiut University
Other Study IDs: ABC
Record Dates: First submitted 2017-08-17; First posted 2017-08-21 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Low Grade group: • 50 tumor tissue samples from patients with Low Grade Bladder Cancer undergoing either trans urethral resection of bladder tumor or Radical Cystectomy ,
  The followings markers must be estimated :
  1. Autophagy markers:
     * ( Atg7) level using (quantitative real time polymerase chain reaction).
     * (LC3A)level using immunohistochemistry .
  2. ER-stress marker: (ATF6) level using ELISA(Enzyme Linked Immuno sorbent Assay)
  3. Oxidative stress Marker:(MDA)using chemical method
  4. Apoptotic marker:(caspase 3) using(quantitative real time polymerase chain reaction) .
- High Grade group: • 50 tumor tissue samples from patients with High Grade Bladder Cancer undergoing either trans urethral resection of bladder tumor or Radical Cystectomy,
  The followings markers must be estimated :
  1. Autophagy markers:
     * ( Atg7) level using (quantitative real time polymerase chain reaction).
     * (LC3A)level using immunohistochemistry .
  2. ER-stress marker: (ATF6) level using ELISA(Enzyme Linked Immuno sorbent Assay)
  3. Oxidative stress Marker:(MDA)using chemical method
  4. Apoptotic marker:(caspase 3) using (quantitative real time polymerase chain reaction) .
- Safety margin group: • 50 normal bladder urothelial tissue samples from the safety margin around the tumor(0.5cm to the tumor),
  The followings markers must be estimated :
  1. Autophagy markers:
     * ( Atg7) level using (quantitative real time polymerase chain reaction).
     * (LC3A)level using immunohistochemistry .
  2. ER-stress marker: (ATF6) level using ELISA(Enzyme Linked Immuno sorbent Assay)
  3. Oxidative stress Marker:(MDA)using chemical method
  4. Apoptotic marker:(caspase 3) using (quantitative real time polymerase chain reaction).
- Control group: • 50 (age and sex matched )control
  The followings markers must be estimated :
  1. Autophagy markers:
     * ( Atg7) level using (quantitative real time polymerase chain reaction).
     * (LC3A)level using immunohistochemistry .
  2. ER-stress marker: (ATF6) level using ELISA(Enzyme Linked Immuno sorbent Assay)
  3. Oxidative stress Marker:(MDA)using chemical method
  4. Apoptotic marker:(caspase 3) using (quantitative real time polymerase chain reaction)..

SUMMARY:
• Bladder cancer is the most common malignancy of the urinary tract. It represents the 7th most commonly diagnosed cancer in male population worldwide and drops to the 11th when both genders are considered . According to the American cancer society's estimates of bladder cancer in 2017, the number of the new cases of bladder cancer is 79,030, and the mortality figures reached 16,870 .

DETAILED DESCRIPTION:
* In Egypt, Bladder Cancer is the most prevalent malignancy among Egyptian males (16%) producing more than 7900 deaths annually . The majority of patients with bladder cancer about (70-80%) present with non-muscle invasive bladder cancer .
* Autophagy is a highly conserved catabolic process that degrades cellular organelles and proteins to maintain cellular biosynthesis during stress ; cancer cells induced autophagy to counteract with anticancer therapy by helping them to evade apoptotic pathway .Autophagy is achieved by many autophagy-related genes .
* Previous studies found that human bladder cancer cell lines exhibit high basal level of autophagic activity that may contribute to resistance to current anticancer treatment, so targeting basal autophagy may help to develop novel therapeutic strategies . Autophagy is potently induced by activating transcription factor 6(Endoplasmic Reticulum stress marker) , and Malondialdehyde (oxidative stress marker) .
* Recently several studies demonstrated the role of autophagy in Bladder Cancer progression as evidenced by detection of microtubule associated protein and its relevance with muscle invasion beside its grade dependency . Autophagy was grade dependent process . Autophagy related gene 7 is a key protein involved in autophagosomes biogenesis, Knockdown of Autophagy related gene 7 induced apoptotic cell death in bladder cancer cell lines measured by increased caspase 3 level, Based on these previous studies autophagy plays a role in bladder cancer progression so interruption of its pathway may serve a novel target for future therapies.

ELIGIBILITY:
Inclusion Criteria:

* 1)patients confirmed histopathologically to have bladder cancer. 2) Both sexes. 3) Patients who will accept to participate in the study.

Exclusion Criteria:

* Patients with past history of Bladder Cancer with previous chemotherapy or any other types of cancer in the last 5 years.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with confirmed bladder cancer (histopathologically) having LGBC(Low Grade bladder cancer) undergoing either TUR(transurethral resection of Bladder Tumour) or Radical Cystectomy and patients having HGBC(High Grade bladder cancer) undergoing either TUR(transurethral resection of Bladder Tumour) or Radical cystectomy. Healthy controls[age and gender matched](with no previous history of gross hematuria, urolithiasis, or active urinary tract infection)
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2021-10-01 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
autophagy marker | baseline
  differences in the level of Atg7(autophagy marker) in Low Grade bladder cancer and High Grade bladder cancer groups in comparison with safety margin and healthy control group.

SECONDARY OUTCOMES:
stress markers | baseline
  Relation between LC3A and muscle invasiveness in bladder cancer progression, and relation between levels of ATF6, activating transcription factor6 (ER stress marker) -MDA malondialdehyde (oxidative stress marker)-Caspase3 (apoptotic marker) in different study groups and bladder cancer development.

CONTACTS AND LOCATIONS:
Overall Officials: Shaimaa Shakhoun, Principal Investigator — Assiut
Locations (1):
- Assiut, Asyut, Egypt

REFERENCES:
- [Result] Woldu SL, Bagrodia A, Lotan Y. Guideline of guidelines: non-muscle-invasive bladder cancer. BJU Int. 2017 Mar;119(3):371-380. doi: 10.1111/bju.13760. Epub 2017 Jan 24. PMID 28058776
- [Result] Mathew R, Karantza-Wadsworth V, White E. Assessing metabolic stress and autophagy status in epithelial tumors. Methods Enzymol. 2009;453:53-81. doi: 10.1016/S0076-6879(08)04004-4. PMID 19216902
- [Result] Kondo Y, Kanzawa T, Sawaya R, Kondo S. The role of autophagy in cancer development and response to therapy. Nat Rev Cancer. 2005 Sep;5(9):726-34. doi: 10.1038/nrc1692. PMID 16148885
- [Result] Mizushima N. Autophagy: process and function. Genes Dev. 2007 Nov 15;21(22):2861-73. doi: 10.1101/gad.1599207. PMID 18006683
- [Result] Lin YC, Lin JF, Wen SI, Yang SC, Tsai TF, Chen HE, Chou KY, Hwang TI. Inhibition of High Basal Level of Autophagy Induces Apoptosis in Human Bladder Cancer Cells. J Urol. 2016 Apr;195(4 Pt 1):1126-35. doi: 10.1016/j.juro.2015.10.128. Epub 2015 Oct 28. PMID 26519656
- [Result] Maiuri MC, Zalckvar E, Kimchi A, Kroemer G. Self-eating and self-killing: crosstalk between autophagy and apoptosis. Nat Rev Mol Cell Biol. 2007 Sep;8(9):741-52. doi: 10.1038/nrm2239. PMID 17717517
- [Result] Yang ZJ, Chee CE, Huang S, Sinicrope FA. The role of autophagy in cancer: therapeutic implications. Mol Cancer Ther. 2011 Sep;10(9):1533-41. doi: 10.1158/1535-7163.MCT-11-0047. Epub 2011 Aug 30. PMID 21878654
- [Result] Sivridis E, Koukourakis MI, Mendrinos SE, Touloupidis S, Giatromanolaki A. Patterns of autophagy in urothelial cell carcinomas--the significance of "stone-like" structures (SLS) in transurethral resection biopsies. Urol Oncol. 2013 Oct;31(7):1254-60. doi: 10.1016/j.urolonc.2011.12.016. Epub 2012 Jan 24. PMID 22281431
- [Result] Ojha R, Singh SK, Bhattacharyya S, Dhanda RS, Rakha A, Mandal AK, Jha V. Inhibition of grade dependent autophagy in urothelial carcinoma increases cell death under nutritional limiting condition and potentiates the cytotoxicity of chemotherapeutic agent. J Urol. 2014 Jun;191(6):1889-98. doi: 10.1016/j.juro.2014.01.006. Epub 2014 Jan 15. PMID 24440234
- [Result] Mukhopadhyay S, Sinha N, Das DN, Panda PK, Naik PP, Bhutia SK. Clinical relevance of autophagic therapy in cancer: Investigating the current trends, challenges, and future prospects. Crit Rev Clin Lab Sci. 2016 Aug;53(4):228-52. doi: 10.3109/10408363.2015.1135103. Epub 2016 Feb 16. PMID 26743568